CLINICAL TRIAL: NCT03393897
Title: Respiratory Variations of the Diameter of Superior Vena Cava for Predicting Fluid Responsiveness After Cardiac Surgery
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Responsible Party: Sponsor
Other Study IDs: IRBN662017
Record Dates: First submitted 2018-01-03; First posted 2018-01-09 (Actual); Last update posted 2018-12-19 (Actual); Status verified 2018-01

CONDITIONS: Transesophageal Echocardiography; Vena Cava Superior
Keywords: fluid responsiveness; cardiac surgery

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Hemodynamic instability with hypotension
  Interventions: Other: Trans oesophageal echocardiography; Other: Trendelenburg test

INTERVENTIONS:
Other: Trans oesophageal echocardiography — Transoesophageal echocardiography : it's a standard practice for this patient
Other: Trendelenburg test — Trendelenburg test : it's a standard practice for this patient

SUMMARY:
In a recent study (Vignon 2017), respiratory variations of the diameter of superior vena cava had a greater diagnostic accuracy than pulse pressure variations and inferior vena cava respiratory variations in 540 medical and surgical ICU patients. But this indicator has not been investigated yet in cardiac surgery. The investigator aim to study respiratory variations of superior vena cava for predicting fluid responsiveness after cardiac surgery.

In post-operative cardiac surgery patients with hemodynamic failure, the investigator will measure respiratory vena caval variations with TEE (Trans oesophageal echocardiography). Then, the investigator will evaluate fluid responsiveness after a fluid challenge (Trendelenburg).

A ROC curve will be constructed in order to assess the optimal sensitivity and specificity of this parameter.

ELIGIBILITY:
Inclusion Criteria:

* Hemodynamic instability with hypotension,
* Low cardiac output or norepinephrine requirements in the first 6 post-operative hours.

Exclusion Criteria:

* TEE (Trans oesophageal echocardiography) contra-indication
* Trendelenburg contra-indication

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with hemodynamic instability and hypotension
Sampling Method: Non-Probability Sample
Enrollment: 56 (Actual)
Dates: Start 2018-01-03 (Actual); Primary Completion 2018-10-31 (Actual); Study Completion 2018-10-31 (Actual)

PRIMARY OUTCOMES:
diameter of vena cava superior | at 6 post-operative hours
  measured with trans oesophageal echocardiography

SECONDARY OUTCOMES:
% of respiratory variations of maximal Doppler velocity in left ventricular outflow tract | at 6 post-operative hours
  measured with trans oesophageal echocardiography
% of respiratory variations of maximal Doppler velocity in pulmonary artery | at 6 post-operative hours
  measured with trans oesophageal echocardiography
% of pulse pressure respiratory variations | at 6 post-operative hours
  measured with trans oesophageal echocardiography

CONTACTS AND LOCATIONS:
Overall Officials: Olivier PEYROUSET, MD, Principal Investigator — CHU SAINT-ETIENNE
Locations (1):
- Centre Hospitalier Universitaire de Saint Etienne, Saint-Etienne, France

IPD SHARING:
Plan to Share IPD: No